CLINICAL TRIAL: NCT01076608
Title: Diabetes Cardiovascular Risk-Evaluation: Targets and Essential Data for Commitment of Treatment (DETECT)
Brief Title: DETECT-Diabetes Cardiovascular Risk-Evaluation: Targets and Essential Data for Commitment of Treatment
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other); Max-Planck-Institute of Psychiatry (Other); University of Magdeburg (Other); Medical University of Graz (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Prof. Dr. H-U.Wittchen, Institute for Clinical Psychology and Psychotherapy, Technical University of Dresden, Germany
Other Study IDs: 149092003
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Cardiovascular Diseases
Keywords: primary care patients
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular diseases are, along with cancer, the most frequent causes for mortality and morbidity in the industrialized nations. Numerous clinical efficient approaches to reduce the known risk factors have been introduced in clinical routine care; yet with quite limited success, e.g. modification of behavioral risk factors, drug treatment and the combination of both. On the population level only marginal changes have been demonstrated, i.e. the mortality from myocardial infarction and stroke remains high.

To answer questions about underlying factors, for this unsatisfactory status, we might profit tremendously from studies that examine the situation, where treatment of patients most frequently take place: in primary care. This approach pays attention to the General Practitioner's (GP) in their gate keeping function in health care. Information from primary care in particular is largely lacking as recently stated by the "Sachverständigenrat für die konzertierte Aktion im Gesundheitswesen" in 2001. The DETECT study has been designed to address these critical issues.

On 16th and 18th September 2003, 3,188 GPs completed a standardised assessment of the diagnostic and therapeutic profile of 55,518 unselected consecutive patients. All patients completed a questionnaire on their demographic data, their complaints, their illness history, their knowledge about selected diseases and their attitude towards those. A sub sample of 7,519 patients additionally attended a standardized laboratory screening program. In this screening the focus was on blood constituents connected with cardiovascular diseases and diabetes, including e. g. cholesterol, lipoproteins, triglycerides and HbA1c. These patients were assessed a second time in the follow up period after one year in 2004 and for a final time after completion of the five-year follow-up period.

DETAILED DESCRIPTION:
What kind of information will DETECT provide?

I. From the cross sectional part (descriptive epidemiological part on 16th/18th September 2003)

* Frequency, characteristics and severity of cardiovascular diseases, selected associated metabolic syndromes and atherosclerotic diseases and syndromes
* Identification and determination of the proportion of patients with high-risk constellations (e.g., post myocardial infarction, associated morbidities, laboratory measures)
* Rates of General Practitioners recognition, diagnostic and therapeutic profiles
* Assessment of quality of care (comparison with guidelines)
* Indicators of undertreatment, overtreatment and inadequate treatment

II. From the longitudinal part

Changes of laboratory parameters and diagnoses after one and five years, in relation to:

* Initial diagnostic and therapeutic status
* Selected intervention criteria
* Composition of risk indicators, and comparison with existing indices (PROCAM, Framingham, Score etc.)
* Measurement of frequency and point of critical outcomes e.g., myocardial infarction, associated morbidity, hospitalisation, critical medical interventions
* Significance of established and "new" cardiovascular risk factors
* Prognostic value of biomarkers for risk stratification

ELIGIBILITY:
Inclusion Criteria:

* unselected primary care patients

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative random sample of 3188 General Practitioners in Germany (general practitioners and internists serving as GPs), who included patients:
  * Main study: 55,518 (unselected consecutive)
  * Longitudinal observation study in a random subset of 7519 patients
Sampling Method: Probability Sample
Enrollment: 55518 (Actual)
Dates: Start 2003-09; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Ullrich Wittchen, Prof. Dr., Principal Investigator — Director of the Institute of Clinical Psychology and Psychotherapy at the Technical University of Dresden

REFERENCES:
- [Background] Wittchen HU, Glaesmer H, Marz W, Stalla G, Lehnert H, Zeiher AM, Silber S, Koch U, Bohler S, Pittrow D, Ruf G; DETECT-Study Group. Cardiovascular risk factors in primary care: methods and baseline prevalence rates--the DETECT program. Curr Med Res Opin. 2005 Apr;21(4):619-30. doi: 10.1185/030079905X38187. PMID 15899112
- See also: Study homepage — http://www.detect-studie.de/index_e.html